CLINICAL TRIAL: NCT00621543
Title: Insertion of an IUD After Medical Abortion
Brief Title: Insertion of an Intrauterine Device (IUD) After Medical Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: University of Utah (Other)
Responsible Party: Dr. Sarah J. Betstadt, Boston University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-24902; H-24902
Record Dates: First submitted 2008-01-28; First posted 2008-02-22 (Estimated); Results first posted 2011-07-08 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: Intrauterine Device Expulsion; Medical Abortion; Induced Abortion
Keywords: Intrauterine Device; Induced Abortion; Medical Abortion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Observation- All subjects (Experimental): Women choosing intra-uterine contraception after medical abortion.
  Interventions: Device: IUD insertion [Copper T-380A or Levonorgestrel (intrauterine system) IUS]

INTERVENTIONS:
Device: IUD insertion [Copper T-380A or Levonorgestrel (intrauterine system) IUS] — When a subject has chosen a method of intra-uterine contraception and has agreed to participate in the study, she will have the intra-uterine device of her choice inserted according to the Food and Druga Administration (FDA) instructions.
  Other Names: IUD insertion icludes the insertion of either the Copper T-380A or Levonorgestrel (intrauterine system) IUS

SUMMARY:
The purpose of this study is to determine the expulsion and continuation rate of an intruterine device (IUD) placed immediately after medical abortion.

Our hypothesis is that immediate-placement of an IUD after completed medical abortion will have a similar expulsion and continuation rate to traditional placement (4-6 weeks after pregnancy).

DETAILED DESCRIPTION:
Women who seek abortion care often desire more effective or longer- lasting contraception. Intrauterine devices are as efficacious as tubal ligation, require no on-going effort on the woman's part to protect her from pregnancy, and are underutilized in the US. We are interested in determining whether placement of an intreatuereine device (IUD) at the time of confirming the completion of a medical abortion may have similar expulsion and continuation rates as IUDs placed after pregnancy (usually a 4-6 week time period). If this is the case, women may save the time and effort of yet another clinic visit, as well as have immediate protection against pregnancy after their abortion. FDA labeling does not specify or restrict time of insertion and therefore this study is in compliance with FDA labeling.

ELIGIBILITY:
Inclusion Criteria:

* Women who completed a medical abortion in the last 14 days
* At least 18 years old.
* Desiring long-term contraception with an IUD.
* Able and willing to give consent for participation in research.
* Gonorrhea and chlamydia screen negative within 60 days of entry to study.
* Willing to comply with the study requirements.
* Accessible by telephone.

Exclusion Criteria:

* Had pelvic inflammatory disease or a septic abortion within the past 3 months or gonorrheal or chlamydial infection in the last 60 days.
* Allergy to copper, or Wilson's disease (for Paragard; may have Mirena)
* Intracavitary of symptomatic uterine fibroids.
* Ovarian, cervical or endometrial cancer.
* Severe anemia (defined as hgb < 8).

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2006-03; Primary Completion 2008-05 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah J Betstadt, MD, Principal Investigator — Boston University; Lynn Borgatta, MD, MPH, Study Director — Boston University
Locations (2):
- United States (2):
  - Boston Medical Center, Boston, Massachusetts
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Background] Henshaw SK, Kost K. Abortion patients in 1994-1995: characteristics and contraceptive use. Fam Plann Perspect. 1996 Jul-Aug;28(4):140-7, 158. PMID 8853278
- [Background] Hubacher D, Cheng D. Intrauterine devices and reproductive health: American women in feast and famine. Contraception. 2004 Jun;69(6):437-46. doi: 10.1016/j.contraception.2004.01.009. PMID 15157788
- [Background] Kaunitz AM. Beyond the pill: new data and options in hormonal and intrauterine contraception. Am J Obstet Gynecol. 2005 Apr;192(4):998-1004. doi: 10.1016/j.ajog.2004.12.091. PMID 15846172
- [Background] Hubacher D, Lara-Ricalde R, Taylor DJ, Guerra-Infante F, Guzman-Rodriguez R. Use of copper intrauterine devices and the risk of tubal infertility among nulligravid women. N Engl J Med. 2001 Aug 23;345(8):561-7. doi: 10.1056/NEJMoa010438. PMID 11529209
- [Background] Penney G, Brechin S, de Souza A, Bankowska U, Belfield T, Gormley M, Olliver M, Hampton N, Howlett-Shipley R, Hughes S, Mack N, O'Brien P, Rowlands S, Trewinnard K; Faculty of Family Planning and Reproductive Health Care Clinical Effectiveness Unit. FFPRHC Guidance (January 2004). The copper intrauterine device as long-term contraception. J Fam Plann Reprod Health Care. 2004 Jan;30(1):29-41; quiz 42. doi: 10.1783/147118904322701956. PMID 15006311
- [Background] El-Tagy A, Sakr E, Sokal DC, Issa AH. Safety and acceptability of post-abortal IUD insertion and the importance of counseling. Contraception. 2003 Mar;67(3):229-34. doi: 10.1016/s0010-7824(02)00518-8. PMID 12618259
- [Background] Stanwood NL, Grimes DA, Schulz KF. Insertion of an intrauterine contraceptive device after induced or spontaneous abortion: a review of the evidence. BJOG. 2001 Nov;108(11):1168-73. doi: 10.1111/j.1471-0528.2003.00264.x. PMID 11762657
- [Background] Christin-Maitre S, Bouchard P, Spitz IM. Medical termination of pregnancy. N Engl J Med. 2000 Mar 30;342(13):946-56. doi: 10.1056/NEJM200003303421307. PMID 10738054
- See also: Intrauterine Devices. The Mayo Clinic — http://www.bcbsri.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Observation- All Subjects
Started | 120
Completed | 97
Not Completed | 23
Not completed — Lost to Follow-up | 23

BASELINE CHARACTERISTICS:
Arm/Group | Observation- All Subjects
Number analyzed (Participants) | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 120
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 28 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 120

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Women With Expulsion of an Intrauterine Device (IUD) Placed After Medical Abortion.
Time Frame: Three months
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Arm Study
Number analyzed (Participants) | 97
percentage of participants | 4 [0 to 8]

2. Secondary Outcome: Percentage of Women Continuing IUD Use at 3 Months
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Arm Study
Number analyzed (Participants) | 97
percentage of participants | 80. [74 to 86]

ADVERSE EVENTS:
Arm/Group | Observation- All Subjects
Serious Adverse Events (participants affected / at risk) | 0/118
Other Adverse Events (participants affected / at risk) | 0/118

LIMITATIONS AND CAVEATS:
21 women did not return for the 3 months follow-up. Some of the 21 women were contacted earlier 3 months, and none had had an expulsion. 2 women were ineligible at the first visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No